CLINICAL TRIAL: NCT03188406
Title: Gastric Cancer Precursor Lesions (GCPL) Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2020-07070; 17-C-N094; 999917094 (Other: National Cancer Institute)
Record Dates: First submitted 2017-06-14; First posted 2017-06-15 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Intestinal Metaplasia; Gastric Cancer
Keywords: Gastric Intestinal Metaplasia; Epidemiology; Risk stratification; Helicobacter pylori; Precancerous lesions; Gastric atrophy
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gastric tissue, serum, plasma, buffy coat, saliva, urine, and stool.

GROUPS / COHORTS (3):
- Gastric cancer: Patients with clinical or histological diagnosis of stomach cancer
- Gastric intestinal metaplasia: Patients classified as OLGIM >0
- Non-atrophic gastritis: Patients classified as OLGA 0

SUMMARY:
Background:

Gastric cancer is a leading cause of cancer deaths around the world. This disease is a serious problem in places like East Asia, Central and South America, and Eastern Europe. Researchers want to study the causes of gastric cancer and its precursors. They want to reduce the number of people with stomach cancer.

Objectives:

To learn more about bacteria factors and other causes of gastric cancer. To study potential markers associated with precancerous gastric lesions (intestinal metaplasia).

Eligibility:

Adults ages 40-70 years at certain hospitals in Chile who:

Are going to have upper gastrointestinal endoscopies

OR have stomach cancer and need surgery

Design:

Participants will give gastric tissue samples.

Some participants will donate a portion of the stomach tissue that is removed as part of their clinical care.

Participants will give access to reports of their stomach exam. They will allow researchers to photograph the microscope slides of their tissue samples.

Participants will answer questions. The topics of the questions include:

Age, height, weight

Education

Habits including tobacco and alcohol

Personal and family history of disease

Reproductive history

Diet

Some participants will give blood, urine, saliva, and stool samples. Study staff will collect the blood. They will tell the participants how to collect the other samples themselves.

DETAILED DESCRIPTION:
The burden of gastric adenocarcinoma is unevenly distributed, with several Asian and Latin American countries having particularly high incidence rates. Although chronic infection with Helicobacter pylori is the primary cause of this cancer, environmental and host cofactors modify the course of infection and determine whether infected individuals develop cancer. Due to the lack of adequate screening strategies and consequent late diagnosis, trends in mortality are similar to incidence, making this neoplasia the third leading cause of cancer death worldwide. The International Agency for Research on Cancer predicts that there will be no reduction in gastric cancer cases until at least 2030 due to population growth and aging. H. pylori-related gastric carcinogenesis is a multi-step process and mucosal lesions of intestinal metaplasia (IM) and dysplasia confer increased risk of progression. Therefore, case-control studies of these premalignant lesions may provide insights into cancer etiology and inform risk stratification. In addition, biomarkers to identify high-risk individuals are needed for early detection and curative treatment. Accordingly, we propose a 3-year study of Chilean adults undergoing upper gastrointestinal endoscopy for clinical purposes to identify 600 subjects with advanced premalignant lesions (i.e., incomplete-type IM, complete-type IM with extension to gastric corpus and dysplasia) for informative comparisons with 600 controls with non-atrophic gastritis, a benign histologic change apparent in most H. pylori infected individuals. As an additional case group, 100 individuals with newly diagnosed gastric cancer will be recruited from the same clinics. This multidisciplinary project will simultaneously evaluate bacterial, host and environmental factors towards a better understanding of gastric cancer etiology that may guide future efforts for prevention and control. We will explore risk factors that have been insufficiently studied, such as various hormones, H. pylori genomics, non- H. pylori gastric microbiota, and other parasitic infections. We will also evaluate potential noninvasive screening markers, including pepsinogens, hormones, miRNAs and DNA methylation. Results from this study may lead to improved management recommendations for individuals with advanced IM. Additionally, the resulting biobank of gastric tissue, blood, urine, saliva and stool will enable state-of-the-art molecular assays and serve as a resource for future research in this area.

ELIGIBILITY:
* INCLUSION CRITERIA:

Two groups of symptomatic patients aged 40 to 70 years old, who are long term residents of a high gastric cancer risk area:

* Approximately 1300 patients who need upper endoscopy (examination of the lining of the stomach with a flexible tube).
* Approximately 100 patients recently diagnosed with stomach cancer who need surgery as treatment for the disease.

EXCLUSION CRITERIA:

* Pregnant women
* Children

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending gastroenterology services.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Histological diagnosis | At enrollment
  Advanced intestinal metaplasia

CONTACTS AND LOCATIONS:
Overall Officials: M. Constanza Camargo, Ph.D., Principal Investigator — U.S. National Cancer Institute (NCI); Alejandro Corvalan, M.D., Principal Investigator — Pontificia Universidad Catolica (Chile)
Locations (9):
- Chile (9):
  - Universidad de Concepción, Concepción
  - Hospital de Curanilahue, Curanilahue
  - Hospital Intercultural, Nueva Imperial
  - Hospital de Puerto Montt, Port Montt
  - Hospital San Juan de Dios, Santiago
  - Pontificia Universidad Catolica, Santiago
  - Hospital de Temuco, Temuco
  - Hospital de Victoria, Victoria
  - Hospital de Villarrica, Villarrica

REFERENCES:
- [Background] Correa P. Human gastric carcinogenesis: a multistep and multifactorial process--First American Cancer Society Award Lecture on Cancer Epidemiology and Prevention. Cancer Res. 1992 Dec 15;52(24):6735-40. PMID 1458460
- [Background] Gonzalez CA, Sanz-Anquela JM, Gisbert JP, Correa P. Utility of subtyping intestinal metaplasia as marker of gastric cancer risk. A review of the evidence. Int J Cancer. 2013 Sep 1;133(5):1023-32. doi: 10.1002/ijc.28003. Epub 2013 Feb 5. PMID 23280711
- [Background] Bonequi P, Meneses-Gonzalez F, Correa P, Rabkin CS, Camargo MC. Risk factors for gastric cancer in Latin America: a meta-analysis. Cancer Causes Control. 2013 Feb;24(2):217-31. doi: 10.1007/s10552-012-0110-z. Epub 2012 Dec 7. PMID 23224270
- [Background] Capelle LG, de Vries AC, Haringsma J, Ter Borg F, de Vries RA, Bruno MJ, van Dekken H, Meijer J, van Grieken NC, Kuipers EJ. The staging of gastritis with the OLGA system by using intestinal metaplasia as an accurate alternative for atrophic gastritis. Gastrointest Endosc. 2010 Jun;71(7):1150-8. doi: 10.1016/j.gie.2009.12.029. Epub 2010 Apr 9. PMID 20381801
- [Background] Rugge M, Correa P, Di Mario F, El-Omar E, Fiocca R, Geboes K, Genta RM, Graham DY, Hattori T, Malfertheiner P, Nakajima S, Sipponen P, Sung J, Weinstein W, Vieth M. OLGA staging for gastritis: a tutorial. Dig Liver Dis. 2008 Aug;40(8):650-8. doi: 10.1016/j.dld.2008.02.030. PMID 18424244